CLINICAL TRIAL: NCT03913416
Title: Can Pre-operative Flexible 3D Models of Pulmonary Malformations Facilitate Thoracoscopic Resection
Acronym: 3DLP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL19_0030
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Malformation
Keywords: pulmonary malformation; 3D printed models; thoracotomy; thoracoscopy children
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D (Experimental): Surgery with surgeon trained using a 3D printed model of the pulmonary malformation.
  Interventions: Device: 3D printed model
- Control group (Other): Conventional surgery without training using a 3D printed model of the pulmonary malformation.
  Interventions: Other: Control group

INTERVENTIONS:
Device: 3D printed model — Before surgery, the surgeon will have a 3D printed model of the pulmonary malformation as well as the lung, the rib cage and the tracheal trunk based on the initial scanner images. He will then be able to train and plan the surgical strategy, as well as to discuss the pulmonary exclusion with the anesthetist.
  Arms: 3D
Other: Control group — The control group is composed of patients operated with standard surgery
  Arms: Control group

SUMMARY:
The National Rare Diseases plans, the ongoing MALFPULM PHRC and thoracoscopic advents in children, are remarkable improvements in understanding and managing lung malformations. The resection of these malformations is now proposed in most cases to avoid infections which are difficult to treat and to diagnose or to avoid exceptional tumors. Procedures are ideally performed around the age of 5-6 months to take advantage of the lung growth that continues during the first two years of life. The surgical strategies depend of the malformation size, the tumor risk and surgeon choice: conservative surgery with removal of part of the lobe may be preferred over complete resection of the concerned lobe.

If possible, thoracoscopic resection is carried out. The open thoracotomy is more painful and leads to complications such as thoracic deformities, larger scars, blood loss. However, in infants the thoracoscopic work space is small, lung exclusion is challenging and the anatomy (normal or malformative) is difficult to understand in space. The rate of thoracoscopy without conversion to thoracotomy ranges from 98% in one American center with a more radical approach , to 48% in a national cohort. Pulmonary exclusion failure, complexity and size of malformations and intra-operative complications are factors of conversion to thoracotomy . These factors can lead surgeons to perform thoracotomy without attempting thoracoscopy.

3D printing is a thriving research field for its educational or therapeutic potential optimization of management, prosthesis, and organ replacement. 3D printing is particularly adapted to pediatrics, which suffers from the rarity of its pathologies and a large spectrum of size and morphology prohibiting the mass production of models. 3D printing models of complex pulmonary pathologies will allowed for a better anesthetic and surgical approach. The modeling of bronchial, vascular and even parenchymatous anatomy permits a better understanding of the anatomical particularities of each patient. This, in turn, avoids the intra-operative conversions to thoracotomy with a direct benefit for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 1 day to 24 months.
* Patients with pulmonary malformation eligible for surgery
* Parents agreement for surgical treatment
* Parents able to sign an informed consent form
* Patient benefiting from a social insurance system or a similar system

Exclusion Criteria:

* Emergency surgeries (less than 15 days between scanner and surgery)
* Obvious extrapulmonary sequestration on tomographic scanning images
* Patients with other major malformation additionally to pulmonary malformation
* Parents unable to understand the purpose of the trial
* Patient already participating to another clinical trial that might jeopardize the current trial

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
proportion of intent to treat under thoracoscopy vs thoracotomy procedures | Day 1
  Comparisonbetween the 2 groups.

SECONDARY OUTCOMES:
conversion rate from thoracoscopy over thoracoscopy attempted. | Day 1
  Comparison between the 2 groups.
Proportion of effective pulmonary exclusion of the operated lung. | Day 1
Proportion of variation between preoperative and effective strategy | Day 1
  Variation of strategy in terms of type of resection (lobar, sub-lobar or segmental resection)
induction time | Day 1
  Comparison of induction time in minutes between the 2 strategies
Evaluation of pain using EVENDOL scale | Hour 12
  Comparison of pain between the 2 groups. Total EVENDOL scores vary from 0 (min) to 15 (max). Each item is scored from 0 to 3 0 = No sign, normal
  1. = weak or transient sign
  2. = moderate or only present half the time
  3. = strong or almost permanent sign
Evaluation of pain using EVENDOL scale | Hour 24
  Comparison of pain between the 2 groups. Total EVENDOL scores vary from 0 (min) to 15 (max). Each item is scored from 0 to 3 0 = No sign, normal
  1. = weak or transient sign
  2. = moderate or only present half the time
  3. = strong or almost permanent sign
Evaluation of pain using EVENDOL scale | Hour 36
  Comparison of pain between the 2 groups. Total EVENDOL scores vary from 0 (min) to 15 (max). Each item is scored from 0 to 3 0 = No sign, normal
  1. = weak or transient sign
  2. = moderate or only present half the time
  3. = strong or almost permanent sign
Evaluation of pain using EVENDOL scale | Hour 48
  Comparison of pain between the 2 groups. Total EVENDOL scores vary from 0 (min) to 15 (max). Each item is scored from 0 to 3 0 = No sign, normal
  1. = weak or transient sign
  2. = moderate or only present half the time
  3. = strong or almost permanent sign
Evaluation of pain using EVENDOL scale | Hour 72
  Comparison of pain between the 2 groups. Total EVENDOL scores vary from 0 (min) to 15 (max). Each item is scored from 0 to 3 0 = No sign, normal
  1. = weak or transient sign
  2. = moderate or only present half the time
  3. = strong or almost permanent sign
percentage of analgesic treatments | Day 10
  Comparison of Analgesic consumption between the 2 groups
Blood loss | Day 1
  Comparison of Blood loss in ml between the 2 groups
number of residual lesions assessed on TDM scanner images | 1 year
number of complications (duration of postoperative air leak greater than 5 days) | Day 10
number of complications (reoperation) | Day 10
number of complications (pneumothorax). | Day 10
Drainage duration | Day 10
  Comparison between the 2 groups of drainage duration in days (drain removal when loss lower than 50ml)
Length of hospital stay | Day 10
  Comparison between the 2 groups of Length of hospital stay in days
resection complexity classification | Day 10
  Development of a resection complexity classification similar to the PreText classification of hepatoblastoma

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Hameury, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mere Enfant, Bron, France